CLINICAL TRIAL: NCT00048659
Title: YM598 Added to Mitoxantrone/Prednisone to Control Pain in Metastatic Prostate Cancer Patients No Longer Responding to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 598-CL-008
Record Dates: First submitted 2002-11-04; First posted 2002-11-06 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Hormone-Refractory Prostate Cancer; Prostatic Neoplasms
Keywords: Androgen-independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — N-(6-methoxy-5-(2-methoxyphenoxy)-2-(pyrimidin-2-yl)pyrimidin-4-yl)-2-phenylethenesulfonamide

INTERVENTIONS:
Drug: YM598

SUMMARY:
The purpose of this study is to determine if patients who take YM598 in addition to mitoxantrone and prednisone (standard therapy) experience improvement in the pain associated with prostate cancer metastases in the bone.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (14):
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - San Bernardino Urological Associates, San Bernardino, California
  - Western Clinical Research, Inc., Torrance, California
  - Shands Hospital, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Georgia Urology,PA Research Institute, Atlanta, Georgia
  - University of Chicago, Section of Hematology/Oncology, Chicago, Illinois
  - University of Illinois, Department of Urology, Chicago, Illinois
  - Michiana Hematology/Oncology, South Bend, Indiana
  - The Urologic Institute of New Orleans, Gretna, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memphis Cancer Center, Memphis, Tennessee
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (8):
  - Department of Medical Oncology, The Canberra Hospital, Canberra
  - Department of Medical Oncology, Concord Hospital Medical Centre, Concord
  - Division of Oncology Ward, Royal Brisbane Hospital, Herston
  - Department of Clinical Oncology, Royal North Shore Hospital, St Leonards
  - Cancer Care Centre, St. George Hospital, Sydney
  - Department of Medical Oncology, Newcastle Mater Hospital, Waratah
  - Southern Medical Day Care Centre, Wollongong
  - Queen Elizabeth Hospital, Clinical Hematology & Oncology, Woodville
- Belgium (2):
  - Cliniques Universitaires St-Luc, Service d'Urologie, Brussels
  - Centre Hospitalier Notre Dame et Reine Fabiola, Service d'oncologie, Charleroi
- France (4):
  - Centre Paul Papin, Angers
  - Service d'Urologie, Hôpital Henri Mondor, Créteil
  - Pavillon V, Service d'Urologie et de transplatation, Hôpital Edouard Herriot, Lyon
  - Service d' Urologie CHU, Hopital Bichat, Paris
- Germany (4):
  - Krankenhause am Urban, Urologie Dieffenfachstr, Berlin
  - Dept Urology University of Essen, Essen
  - Urologische Klinik der MHH, Hanover
  - Klinikum Mannheim Urology, Mannheim
- Mater Misericordiae Hospital, Dublin, Ireland
- Universitair Medisch Centrum Utrecht, Dienst Medische Oncologie, Utrecht, Netherlands
- Poland (7):
  - Kilinika Chemioterapii, Centrum Onkologii Instytut im M sklodowskiej Curie, Krakow
  - Oddzial Chemioterapii, Krakow
  - Klinika Chemioterapii AM, Lodz
  - Samodzielny Publiczny Zaklad Opieki zdrowotnej, Wojewodzki Osrodek Onkologii, Opole
  - Szpital Wojewodzki im Sw Lukasza SP ZOZ Tarnow, Tarnów
  - Klinika Nowotworow Ukladu, Warsaw
  - Szpital CSK WAMl, Klinika Okologii, Warsaw
- Spain (5):
  - Hospital Clinic i Provincial, Servicio de Oncologia, Barcelona
  - Hospital General Vall d'Hebron, Servicio de Oncología, Barcelona
  - Hospital Universitario de Getafe, Servicio de Urologia, Crta, Getafe (Madrid)
  - Hospital Universitario Príncipe de Asturias, Servicio de Urología, Madrid
  - Instituto Valenciano de Oncologia, Servicio de Oncologia, Valencia
- United Kingdom (7):
  - Department of Urological Research, Derriford Hospital, Devon
  - Clinical Research Centre, St George's Hospital, Urology Division, London
  - Department of Urology, St Bartholomew's Hospital, London
  - Imperial College School of Medicine, Dept Cancer Medicine, London
  - Department of Urology, East Surrey Hospital, Surrey
  - Royal Surrey County Hospital, Surrey
  - St Richard's Hospital, West Sussex